CLINICAL TRIAL: NCT05175612
Title: Differentiation of Upper and Lower Respiratory Tract Infections Using Automated Lung Sound Analysis With LungPass Device
Status: Suspended | Type: Observational
Why Stopped: For sponsor reasons
Sponsor: Healthy Networks (Industry)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: № 4-3/YH-2056/LP06
Record Dates: First submitted 2021-11-26; First posted 2022-01-04 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Tract Infection
Keywords: Lung sound analysis; Upper Respiratory Truct Infections; Lower Respiratory Truct Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lung auscultation with LungPass device (electronic auscultation) — Lung auscultation with electronic stethoscope

SUMMARY:
This observational study evaluates whether lung sound analysis with LungPass device can be used to differentiate upper and lower respiratory tract infections (URTI and LRTI)

DETAILED DESCRIPTION:
This is a prospective observational study comprised patients presenting with acute respiratory tract infection symptoms in primary care settings. Patients will undergo routine clinical examination including lung auscultation with conventional stethoscope and LungPass device. Moreover, symptoms and anamnesis data, result of diagnostic questionnaire from the LungPass App, complete blood count, C-reactive protein, procalcitonin (PCT) level, SARS-CoV-2 PCR test and X-ray chest examination or CT chest (in case of preliminary clinical suspicion of LRTI). Patients will be followed up within 5-7 days and at the end of the disease in person or by phone for clinical course of the disease assessment to confirm the final diagnosis (URTI or LRTI). Final diagnosis will be considered as Gold standard for accuracy assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years) and children (3-18 years) of both sexes;
* Patients able and willing to sign an informed consent to participate in the study (parents of children younger than 18 years old will be allowed to give an informed consent on behalf of their children).
* Patients presenting with a new onset of at least two of listed acute respiratory tract infection symptoms within the last 5 days: cough, purulent sputum, breathlessness, core temperature above 38°C.
* Patients who first visit a GP with these symptoms within the first 5 days from the onset of symptoms and was not previously treated with antibiotics during the last month.

Exclusion Criteria:

* Age up to 3 years;
* Patient refusal to participate in the study (or patients' parents);
* Children under full State care (orphans, children left without parental care);
* Treatment with antibiotics during the last month;
* Patients with subcutaneous emphysema, with damaged skin on the surface of the chest, with drainage in the pleural space, patients undergoing mechanical ventilation;
* Presence of other known chronic lung conditions such as asthma, COPD, tuberculosis, cystic fibrosis or bronchiectasis;
* Mental illness, other known acute diseases or known chronic decompensated diseases, such as a known active malignancy or severe heart failure.
* Other known ongoing infection.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited in primary care settings upon presentation with symptoms of acute respiratory infection.
  It is planned to start recruiting 100 adult patients and 100 children with URTI and 100 adults and 100 children with LRTI. The final calculation of the sample size will be carried out after receiving the preliminary results of the study. After that, the sample size will be adjusted.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of identifying LRTI by abnormal lung sounds | 16.11.2021- 30.11.2021
  Accuracy of differentiation between ULRTI and LRTI by abnormal lung sounds detected with LungPass device

SECONDARY OUTCOMES:
Accuracy of identifying LRTI by abnormal lung sounds in subgroups with COVID-19 and non-COVID-19 LRTI | 16.11.2021- 30.11.2021
  Accuracy of differentiation between ULRTI and LRTI by abnormal lung sounds detected with LungPass device in subgroups with COVID-19 and non-COVID-19 LRTI
Lung sounds and clinical signs of LRTI correlation in patients with LRTI | 16.11.2021- 30.11.2021
  Correlation between presence of pathological pulmonary sounds detected with LungPass device and presence of clinical signs of LRTI (clinical parameters/radiology results) in patients with LRTI

OTHER OUTCOMES:
Accuracy of LRTI detection by LungPass App output | 16.11.2021- 30.11.2021
  Accuracy of of identifying LRTI by LungPass App output which based on abnormal lung sounds detected with LungPass device together with symptoms collected using a questionnaire in the LungPass app*.
  * Final LungPass App output is possible patient condition (acute respiratory infection, acute bronchitis, pneumonia, etc)
Accuracy of bacterial LRTI detection by abnormal lung sounds using procalcitonin level as Gold Standard | 16.11.2021- 30.11.2021
  Accuracy of identifying bacterial LRTI by abnormal lung sounds detected with LungPass device using procalcitonin level as Gold Standard

CONTACTS AND LOCATIONS:
Overall Officials: Helena Binetskaya, Study Director — CEO
Locations (1):
- 19th Сentral District Polyclinic of Pervomaisky District of Minsk, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided